CLINICAL TRIAL: NCT01395173
Title: Position Changes During Colonoscope Withdrawal to Increase Polyp Detection: a Prospective Randomized Trial
Brief Title: Position Changes During Colonoscope Withdrawal and Polyp Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H11-00087
Record Dates: First submitted 2011-07-13; First posted 2011-07-15 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Colonic Polyp
Keywords: detection
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Subject will undergo standard colonoscopy.
  Interventions: Procedure: Standard
- Position change (Active Comparator): Subject will under go standard colonoscopy, but also with position changes during colonoscope withdrawal.
  Interventions: Procedure: Position change

INTERVENTIONS:
Procedure: Position change — Patients will be randomly assigned to two groups: Control group (those who will receive standard colonoscopy without position changes) and Position change group (those who will undergo position changes during colonoscope withdrawal during colonoscopy). Subjects in position change group will be asked to shift into three different positions during colonoscope withdrawal.
  Arms: Position change
Procedure: Standard — Subjects will undergo standard colonoscopy without position changes during scope withdrawal.
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether position changes during colonoscope withdrawal affects polyp detection rate. We hypothesize that positions change during scope withdrawal will increase polyp detection rate.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients undergoing colonoscopy
* Age 40 or greater

Exclusion Criteria:

* Inpatient colonoscopy
* Unable to provide informed consent
* Unable to complete colonoscopy to cecum
* Previous bowel resection, inflammatory bowel disease, polyposis syndrome
* Musculoskeletal disorder or other mobility issue limiting effective patient position changes
* Inadequate bowel preparation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 776 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Polyp detection rate | 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Telford, MD, FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Ou G, Kim E, Lakzadeh P, Tong J, Enns R, Ramji A, Whittaker S, Ko HH, Bressler B, Halparin L, Lam E, Amar J, Telford J. A randomized controlled trial assessing the effect of prescribed patient position changes during colonoscope withdrawal on adenoma detection. Gastrointest Endosc. 2014 Aug;80(2):277-83. doi: 10.1016/j.gie.2014.01.032. Epub 2014 Mar 12. PMID 24629419